CLINICAL TRIAL: NCT02651818
Title: The Impact of Surgical Treatment of Benign Non-toxic Goiter on Quality of Life
Brief Title: Changes in Quality of Life Following Surgical Treatment of Benign Non-toxic Goiter
Acronym: SOLOIST
Status: Completed | Type: Observational
Sponsor: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Jesper Roed Sorensen, MD, University of Southern Denmark
Other Study IDs: S-20132
Record Dates: First submitted 2016-01-06; First posted 2016-01-11 (Estimated); Last update posted 2018-05-15 (Actual); Status verified 2018-05

CONDITIONS: Goiter
Keywords: Goiter; Thyroid disease; Struma
MeSH Terms: conditions — Goiter; Thyroid Diseases | interventions — Thyroidectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Thyroidectomy — Regular thyroidectomy or hemithyroidectomy through Kocher's skin incision

SUMMARY:
The aim is to investigate the influence of surgical treatment on benign non-toxic goiter on the disease specific quality of life evaluated 6 months after thyroid surgery.

All investigations follow already scheduled treatments.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing hemi- or total thyroidectomy for benign non-toxic goiter with pressure symptoms
* The patients must be able to understand, read and write Danish

Exclusion Criteria:

* Previous surgery to the neck
* Diabetes or any neuromuscular disorders
* Present or previous head and neck malignancy, including malignancy found in the surgical thyroid specimen or suspicion hereof

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing hemi- or total thyroidectomy at Odense University Hospital for benign symptomatic non-toxic goiter
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2014-10-30 (Actual); Primary Completion 2017-10-24 (Actual); Study Completion 2017-10-24 (Actual)

PRIMARY OUTCOMES:
Change in quality of life following thyroidectomy | 6 months
  Change in goiter symptom score at the Thyroid specific Patient Reported Outcome measure (ThyPRO) following thyroidectomy

CONTACTS AND LOCATIONS:
Overall Officials: Christian Godballe, Professor, Study Director — University of Southern Denmark
Locations (1):
- Odense University Hospital, Odense, Denmark

IPD SHARING:
Plan to Share IPD: Undecided